CLINICAL TRIAL: NCT03053323
Title: Preconception and Pregnancy Obesity Treatment and Prevention Among Women With a History of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Louisa Grandin Sylvia, Director of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002556
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Depression
Keywords: Preconception; Pregnancy; Lifestyle
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lifestyle Intervention (Experimental)
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The lifestyle intervention consists of three components: nutrition, physical activity, and other areas of wellness. The intervention is administered individually each week for 10 weeks and is tailored for women with a history of depression who are in the first trimester of pregnancy or trying to conceive.

SUMMARY:
The purpose of the Preconception and Pregnancy Obesity Treatment and Prevention Among Women with A History of Depression preliminary study is to provide a lifestyle intervention for women with a history of depression who are trying to conceive or are pregnant in order to prevent excessive pre-pregnancy weights, avoid excessive gestational weight gain, and to improve other markers of metabolic health. The treatment program consists of 10 private sessions with a trained clinician at no cost to participants.

DETAILED DESCRIPTION:
The investigators are evaluating a new lifestyle intervention to help women with a history of depression who are pregnant or trying to conceive to learn to exercise, eat well, and live a healthy lifestyle. They are interested in examining if this therapy-based program can positively impact eating and exercising habits and see if the treatment is enjoyable. All participants will receive this intervention.

ELIGIBILITY:
Inclusion Criteria:

* History of depression
* Pregnant in first trimester or planning to become pregnant within next year
* Ability to give informed consent
* Age > or = 18 and < 45 years
* Overweight or obese (Body mass index > 25 kg/m^2)

Exclusion Criteria:

* Unwilling/unable to comply with study procedures
* Endorsed item on the Physical Activity Readiness Questionnaire (PAR-Q)
* Diagnosis of anorexia nervosa or bulimia nervosa in the past month
* Diagnosis of substance dependence in the past month
* Active suicidality (Montgomery Asberg Depression Rating Scale (MADRS) item 10 score > 4)
* Exercising regularly (i.e., 5 days per week for 30 min)
* Neurologic disorder or history of head trauma
* Contraindications to exercise or diet interventions (e.g., co-morbid nutritional and metabolic diseases, physical injuries, contraindications to exercise for pregnant women)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of treatment measured by participation rates | 10 weeks
  Participation rates measure attendance at weekly sessions.
Acceptability of treatment on Client Satisfaction Questionnaire (CSQ-8) | 10 weeks
  The CSQ-8 is a reliable and valid self-report measure of satisfaction with care and perceived quality and acceptability of treatment.

SECONDARY OUTCOMES:
Weight loss | 10 weeks
  Weight will be measured during pre-, mid-, and post-treatment visits.
Exercise duration on the Exercise Questionnaire (EQ) | 10 weeks
  The EQ assesses baseline exercise history and ongoing exercise duration and frequency.
Depression severity on the Montgomery-Asberg Depression Rating Scale (MADRS) | 10 weeks
  The MADRS assesses the presence and severity of patient's current depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Sylvia, PhD, Principal Investigator — Massachusetts General Hospital; Marlene Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No